CLINICAL TRIAL: NCT06727773
Title: Memantine and Exercise to Improve Cognitive Function and Modulate Biological Pathways of Cognitive Decline During Chemotherapy in Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LCCC2425; K23AG086604 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-12-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Locally Advanced Breast Cancer; Cognitive Impairment; Cognitive Decline; Cognitive Change; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
Keywords: chemotherapy; memantine; placebo-controlled; exercise; Get Real & Heel cancer exercise program
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Motor Activity | interventions — Memantine; lime

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to MEM+EX (memantine + exercise), memantine, or placebo using a computer-generated randomization scheme that stratifies for an equal balance of age. All study personnel and participants will remain blinded until data collection is complete.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): Participants will receive study medication (memantine) and Get Real & Heel exercise guided by the therapist.
  Interventions: Drug: Memantine; Other: Exercise Intervention
- Arm 2 (Placebo Comparator): Participants have access to a library of pre-recorded Get Real & Heel sessions.
  Interventions: Drug: Placebo medication; Other: Exercise Control
- Arm 3 (Experimental): Participants will receive study medication (memantine) and access to a library of pre-recorded Get Real & Heel sessions.
  Interventions: Drug: Memantine; Other: Exercise Control

INTERVENTIONS:
Drug: Memantine — memantine capsule
  Arms: Arm 1; Arm 3
Drug: Placebo medication — placebo capsule
  Arms: Arm 2
Other: Exercise Intervention — Exercise Intervention participants will concurrently engage in remotely delivered Get Real & Heel, 3d/week. Intensity for aerobic and strength-training components will progress as tolerated under the direction of a trained exercise physiologist.
  Other Names: Get Real & Heel
  Arms: Arm 1
Other: Exercise Control — Exercise control will have access to a library of pre-recorded Get Real & Heel sessions.
  Other Names: Exercise library
  Arms: Arm 2; Arm 3

SUMMARY:
This randomized, placebo-controlled trial aims to assess the feasibility, acceptability, and preliminary efficacy of memantine and the University of Carolina (UNC)'s Get Real & Heel cancer exercise program (MEM+EX) in addressing cancer-related cognitive impairment (CRCI) and underlying CRCI biomarkers. Ninety stage I-III breast cancer patients with mild cognitive difficulties during chemotherapy will be randomized into three groups: MEM+EX, memantine, or placebo. The study will evaluate recruitment, retention, adherence, acceptability, cognitive function, brain-derived neurotrophic factor (BDNF), inflammatory markers, and frailty at multiple time points.

DETAILED DESCRIPTION:
There are 4 million breast cancer survivors in the U.S. and an estimated 1.4 million suffer from long-term cognitive deficits from cancer treatment. Compared to other cancers and treatments, cognitive decline has been most robustly described in breast cancer and following chemotherapy with up to 75% self-reporting and ~50% objectively demonstrating at least mild cognitive deficits after chemotherapy. Memantine, an N-methyl-D-aspartate receptor antagonist, is a promising medication to address underlying mechanisms of CRCI, including inflammation and pathways involving brain-derived neurotrophic factor (BDNF). Exercise, a promising intervention for frailty which intervenes on multiple mechanisms of aging, is an ideal strategy to augment the targeted effects of memantine.

The primary objective of this study is to demonstrate the feasibility and acceptability of MEM+EX during breast cancer chemotherapy. Secondarily, the preliminary efficacy of MEM+EX and memantine on putative biomarkers of CRCI and cognitive function will be evaluated. Furthermore, the impact of frailty on the preliminary efficacy of MEM+EX and memantine will be explored.

The proposed study has the potential to produce significant public health benefit by filling a major gap in effective CRCI treatments. It will provide important pilot data for future, definitive randomized controlled studies. Finally, this study will advance understanding of potential targets to pursue in future cognitive interventions, including pathways involving BDNF and inflammation, during treatment for cancer.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in the study a subject must meet all of the eligibility criteria outlined below.

* Female
* Age ≥ 50 years at the time of consent.
* Stage I-III Breast Cancer
* Recommended chemotherapy
* Enroll prior to 3rd cycle of chemotherapy
* Completed at least 1 cycle of standard-of-care neoadjuvant or adjuvant chemotherapy
* At least mild self-reported cognitive concerns ≥3 on a 0-10 scale
* English-speaking

Exclusion Criteria:

* Allergy to memantine
* Previous chemotherapy (prior to the current regimen),
* Severe cognitive impairment, defined by Blessed Orientation Memory Concentration Test Score ≥11
* Myocardial infarction in the last 6 months
* Cardiovascular or orthopedic limitations to exercise
* Severe mental illness (i.e., schizophrenia or bipolar affective disorder)
* Current alcohol or drug abuse
* Inability to swallow capsules </= 5mL/min
* CrCl </= 5mL/min

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Rates of recruitment | Baseline
  Rates of recruitment will be measured as a number of subjects joined the study.
Rates of retention | Up to a year
  Rates of retention will be measured as the proportion of subjects who remained in the study at post-intervention (up to 6 months) and after 6 months among those who started the intervention
Rates of adherence | Up to a year
  Rates of adherence will be measured as a number of subjects who joined the study completed 80 percent of planned study activities.
The acceptability of memantine + Get Real and Heel (MEM+EX) | Up to 6 months
  The acceptability of memantine + Get Real and Heel (MEM+EX) will be assessed using the Client Satisfaction Questionnaire (CSQ-3). CSQ-3 is a three-item measure of treatment acceptability that has demonstrated excellent reliability and validity across a range of patient care settings.
  Each item is scored on a Likert-type scale from 1 (low satisfaction) to 4 (high satisfaction). CSQ-3 will be completed at post-intervention only (or at the time of withdrawal from the study, if applicable).

SECONDARY OUTCOMES:
Attention and Executive Function Composite Score | Baseline and up to 1 year
  The attention and executive function score is a composite of the following neuropsychological assessment measures: Digit Span, Trail Making Test Parts A&B, Controlled Oral Word Association Test, and Animal Naming Test. It will be calculated as the sum of Z-scores (standardized based on available age-, sex-, education-, and race/ethnicity-matched normative data) of the individual subtests and range from a Z-score of -3 to +3.
Learning and Memory Composite Score | Baseline and up to 1 year
  The learning and memory score is a composite of the following neuropsychological assessment measures: Hopkins Verbal Learning Test-Revised and Brief Visual Memory Test-Revised. It will be calculated as the sum of Z-scores (standardized based on available age-, sex-, education-, and race/ethnicity-matched normative data) of the individual subtests and range from a Z-score of -3 to +3.
Changes in patient-reported cognition | Baseline and up to 1 year
  The impact of MEM+EX and memantine on cognitive function will be determined by examining changes in patient-reported cognition, as measured by the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog PCI) version 3, compared to placebo.
  FACT-Cog PCI is a self-report measure designed to assess perceived cognitive functioning in cancer patients, particularly those experiencing chemotherapy-induced cognitive problems. It consists of 18 items and each item is rated on a 5-point Likert scale, ranging from 0 (Never) to 4 (Several times a day). The total score is obtained by summing the subscale scores. Higher scores indicate better perceived cognitive functioning.
The impact of MEM+EX and memantine on brain-derived neurotrophic factor (BDNF) | Baseline and up to 6 months
  The impact of MEM+EX and memantine on putative biomarkers of CRCI will be determined by examining changes in BDNF compared to placebo.
The impact of MEM+EX and memantine on inflammatory markers | Baseline and up to 6 months
  The impact of MEM+EX and memantine on putative biomarkers of CRCI will be determined by examining changes in inflammatory composite measure (TNF-alpha, IL-6, CRP) compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Zev Nakamura, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials